CLINICAL TRIAL: NCT05331846
Title: The Effect of Breast Milk Odor on the Pain and Stress Level of the Newborn During the Endotracheal Aspiration Procedure
Brief Title: Breast Milk Odor on the Pain and Stress Level of the Newborn Endotracheal Aspiration Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.O.oı.OO/l 8
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Endotracheal Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMELL OF BREAST MILK (Experimental): the smell of breast milk will reduce pain and stress
  Interventions: Behavioral: the smell of breast milk
- control (No Intervention): pain and stress will not decrease

INTERVENTIONS:
Behavioral: the smell of breast milk — Smell of breast milk during endotracheal aspiration will reduce pain and stress
  Arms: SMELL OF BREAST MILK

SUMMARY:
Our study aims to determine the effect of breast milk odor on pain and stress in the application of endotracheal aspiration in newborns hospitalized in the Neonatal Intensive Care Unit. The research is planned experimentally with a pretest posttest randomized control group. The research will be carried out in Şanlıurfa Training and Research Hospital Neonatal Intensive Care Unit between March-December 2022. The population of the study will consist of patients aged 30-28 days who were hospitalized in the Şanlıurfa Training and Research Hospital Neonatal Intensive Care Unit between March-December 2022 and received mechanical ventilation treatment.

The research sample; Babies of families who are hospitalized on the dates specified with the probability sampling method and meet the research criteria and volunteer to participate in the research will be formed. Questionnaire Form, Neonatal Pain and Stress Assessment Scale, and Follow-up Form will be used to collect research data. The scent of breast milk will be used as an intervention tool in the research.

DETAILED DESCRIPTION:
3.1. Type of Research The research is planned experimentally with a pretest posttest randomized control group.

3.2. Place and Time of Research The research will be carried out in Şanlıurfa Training and Research Hospital Neonatal Intensive Care Unit between March-December 2022.

3.3. Population and Sample of the Research The population of the study will consist of patients aged 30-28 days who were hospitalized in the Şanlıurfa Training and Research Hospital Neonatal Intensive Care Unit between March-December 2022 and received mechanical ventilation treatment.

The research sample; Babies of families who are hospitalized on the dates specified with the probability sampling method and meet the research criteria and volunteer to participate in the research will be formed. In this study, a priori power analysis was performed to determine the sample size. In the power analysis, Cohen's standard effect sizes reference method was chosen. In this case, in our study, for the t-test in independent groups in which the effect of sniffed breast milk on endotracheal aspiration application will be compared, it was determined that "80% power at the 95% confidence interval at the 0.05 significance level" could be reached if the study was conducted with a total of 80 participants in two groups with 40 participants in each group. In case of data loss, it was decided to collect data from a total of 88 individuals by including 10% backup sample to this number. Data will be collected at different times from newborns receiving invasive mechanical ventilation support in incubators in the Neonatal Intensive Care Unit. There is no interaction between the groups.

Inclusion Criteria for Research

* Being a term newborn,
* to be between 0-28 days,
* Receiving mechanical ventilation support,
* Not taking opioids or sedatives 4 hours before the procedure. 3.4. Data Collection Tools to be Used in the Research Questionnaire Form, Neonatal Pain and Stress Assessment Scale, and Follow-up Form will be used to collect research data. The scent of breast milk will be used as an intervention tool in the research.

Questionnaire Form: In this form, which was prepared by the researcher by examining the literature; There will be questions about the introductory features of the newborn.

ALPS Neo Neonatal Pain and Stress Rating Scale: The "Newborn Pain and Stress Rating Scale" was developed in 2014, based on the individualized developmental care of the newborn, in order to assess pain and stress in premature and term newborns. In 2017, this scale was adapted to Turkish and validity and reliability studies were conducted. ALPS Neo "Newborn Pain and Stress Assessment Scale" is a 3-point Likert-type scale consisting of 5 items, including "facial expression, breathing pattern, tone of extremities, hand/foot activities and activity level" of the newborn, and measurements are made by observation. As the scores obtained increase, pain and stress increase in the newborn. As a result of the evaluation, "3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress".

Follow-up Form: It is the form used to record the cardiorespiratory parameters (peak heart rate, oxygen saturation) of the newborn evaluated before, during and after the procedure, ALPS Neo pain scale, and crying time result.

Intervention Tool Used in Research Breast Milk Scent: Breast milk scent will be used as an intervention tool in the research. In the study, breast milk will be sniffed 5 minutes before endotracheal aspiration with the help of sterile sponge. As a non-pharmacological method, it is expected that the smell of breast milk will reduce the pain and stress felt during endotracheal aspiration in the newborn.

3.5. Data Collection The research data will be obtained from the babies of the parents who agreed to participate in the research after the researcher gave the parents of the patients preliminary information about the research (the purpose of the research, why the research was conducted, the attempt to relieve the neonatal pain with a non-pharmacological method, etc.) and their written consent was obtained.

Before the endotracheal aspiration attempt is made by the researcher to the experimental group, the patient will smell the breast milk scent with the help of a sterile sponge for 5 minutes.

The purpose of making the patient smell the breast milk; It is to reduce the pain level of the procedure to the minimum level by ensuring that the patient calms down. The researcher will have the patient smell breast milk for 5 minutes before the endotracheal aspiration procedure and will evaluate the patient with the "ALPS Neo Neonatal Pain and Stress Rating Scale" before, during and after the procedure. The control group will be routinely performed in the endotracheal aspiration procedure and will be evaluated with the "ALPS Neo Neonatal Pain and Stress Rating Scale" before, during and after the procedure.

3.6. Evaluation of Data The processing and statistical analysis of the collected data will be done with the analysis software called SPSS (Statistical Package for the Social Sciences) for Windows 20.0.

3.7. Ethical Principles of Research In order to carry out the research, official permission will be obtained from the relevant institution with ethical approval from the Ethics Committee. The purpose of the study will be explained to the parents of the babies with the research group criteria, the questions asked will be answered and their verbal and written consent will be obtained. Parents will be informed that the data collected during the research will be processed anonymously, confidentially, and will not be used outside of the study in question, and that they can leave the study whenever they wish. Since the research is based on the use of data obtained from humans, and therefore, due to the necessity of observing personal rights, the relevant ethical principles "Informed Consent", "Volunteerism" and "Protection of Confidentiality" will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Being a term newborn,
* to be between 0-28 days,
* Receiving mechanical ventilation support,
* Not taking opioids or sedatives 4 hours before the procedure.

Exclusion Criteria:

* not be between 0-28 days,
* Not receiving mechanical ventilation support,
* Taking opioids or sedatives 4 hours before the procedure.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
ALPS Neo Neonatal Pain and Stress Rating Scale | 9 MONTHS
  In 2014, the "Newborn Pain and Stress Rating Scale" was developed based on the individualized developmental care of the newborn in order to evaluate pain and stress in premature and term newborns. In 2017, this scale was adapted to Turkish and validity and reliability studies were conducted. ALPS Neo "Newborn Pain and Stress Assessment Scale" is a 3-point Likert-type scale consisting of 5 items, including "facial expression, breathing pattern, tone of extremities, hand/foot activities and activity level" of the newborn, and measurements are made by observation. As the scores obtained increase, pain and stress increase in the newborn. As a result of the evaluation, "3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress".

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Study Director — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED